CLINICAL TRIAL: NCT06787703
Title: Are Older Adults Prepared to Respond to Disasters? A Randomized Controlled Study Evaluating the Effectiveness of Psychological First Aid on Dignity-Related Distress, Social Frailty, and Psychological Resilience Among Institutionalized Elders
Brief Title: Are Older Adults Prepared to Respond to Disasters? Psychological First Aid on Dignity-Related Distress, Social Frailty, and Psychological Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Damanhour University (Other); Prince Sattam Bin Abdulaziz University (Other); Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Ahmed Ahmed Elsheikh, Lecturer, Faulty of Nursing, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 106-C
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Elderly; Psychological Adaptation; First Aid; Stress; Psychological Stress
Keywords: Older Adults; Disaster; Psychological; First Aid; Dignity-Related Distress; Psychosocial Frailty; Psychological Resilience; Institutionalized Elders.
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Psychological first aid is a compassionate and supportive presence designed to mitigate acute distress and asses the need for continued mental health care. The intervention aims to enhance the compassionate presence, assist with needs and promote adaptive functioning. The intervention encompasses seven main themes (RAPID model, emotion stabilization, self-compassion, reframing, instillation of hope and empowerment) that will be covered through a series of five training exercises conducted on 6 sessions. Each session ranged in duration from 30 to 45 minutes.
Masking Description: NO masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): standard care
- Psychological First Aid Intervention (Experimental): Psychological First Aid Intervention
  Interventions: Behavioral: Psychological First Aid Intervention

INTERVENTIONS:
Behavioral: Psychological First Aid Intervention — Psychological first aid is a compassionate and supportive presence designed to mitigate acute distress and asses the need for continued mental health care. The intervention aims to enhance the compassionate presence, assist with needs and promote adaptive functioning. The intervention encompasses seven main themes (RAPID model, emotion stabilization, self-compassion, reframing, instillation of hope and empowerment) that will be covered through a series of five training exercises conducted on 6 sessions. Each session ranged in duration from 30 to 45 minutes.
  The program going along the RAPID PFA model, that represents a simple structure of (R for: establishing rapport and reflective listening, A: assessment, P: prioritization, I: intervention and D: disposition).
  The program going along the RAPID PFA model, that represents a simple structure of (R for: establishing rapport and reflective listening, A: assessment, P: prioritization, I: intervention and D: disposition). The
  Arms: Psychological First Aid Intervention

SUMMARY:
The rapid increase in the global aging population has drawn attention to the unique challenges faced by institutionalized elders. These individuals often contend with various forms of psychosocial stress, including dignity-related distress, social frailty, and reduced psychological resilience. Dignity-related distress, characterized by feelings of worthlessness or loss of respect, significantly impacts mental health and quality of life among older adults, especially those in long-term care facilities. Similarly, social frailty-marked by diminished social networks and weakened interpersonal interactions-further exacerbates their vulnerability to loneliness and mental health disorders. Enhancing psychological resilience, or the capacity to adapt to adversity, is therefore critical to improving their overall well-being.

Psychological First Aid (PFA) is a structured intervention designed to provide immediate support and foster adaptive coping strategies during crises. While PFA has been widely implemented in disaster and emergency contexts, its application in addressing the psychosocial needs of institutionalized elders remains underexplored. Given its focus on promoting safety, comfort, and connectedness, PFA may hold potential for mitigating dignity-related distress, strengthening social bonds, and enhancing psychological resilience among this vulnerable population.

This study seeks to evaluate the effectiveness of PFA in alleviating dignity-related distress, reducing social frailty, and bolstering psychological resilience among institutionalized elders. By addressing these intertwined psychosocial factors, the research aims to contribute to the growing body of evidence on interventions tailored to the unique needs of older adults in care settings

DETAILED DESCRIPTION:
The study addresses critical aspects of elderly care, particularly for those in institutional settings. Institutionalized elders often face challenges such as diminished dignity, social isolation, and reduced resilience, which can significantly impact their mental and emotional well-being. By evaluating the role of Psychological First Aid (PFA), a practical and empathetic intervention designed to provide immediate emotional support, the study explores its potential to alleviate dignity-related distress, mitigate social frailty, and enhance psychological resilience. The findings have important implications for improving the quality of life for institutionalized elders by promoting a sense of self-worth, strengthening social connections, and fostering adaptability to life's challenges, ultimately contributing to a more holistic approach to elder care.As well, this study involved an innovative application of the psychological first aid interventions. While PFA has been widely used in disaster response and emergency settings, its application in addressing the day-to-day struggles of institutionalized elders is novel. The study expands the scope of PFA, demonstrating its adaptability and potential for broader usage in healthcare and social care settings. The findings of this study could influence policies and practices in eldercare by advocating for the integration of PFA into standard care protocols. It highlights the need for training caregivers in PFA to improve the holistic care of institutionalized elders. In general, the study adds to the growing body of gerontological research, offering evidence-based strategies to address the complex psychological and social needs of the aging population in institutional settings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older.
* Recently retired, within a maximum of one month from job cessation.
* Capable of meaningful and clear communication.
* Provide signed informed consent to participate.

Exclusion Criteria:

* Participation in psychological treatments
* Inability to complete assigned homework
* Unwillingness to continue studying
* Logistical challenges such as poor internet connectivity during online sessions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Psychological Resilience Evaluation Scale | at baseline assessment before the start of the program and at 3 months immediately after the completion of the study
  The Resilience Evaluation Scale (RES) consists of 9 items rated on a 5-point Likert scale ranging from 0 (completely disagree) to 4 (completely agree). Participants assess the extent to which they agree with statements about how they "typically respond to challenging situations." the scale's original authors identified a two-factor structure: self-efficacy, which includes items 2, 3, 4, 5, 6, and 8 (subscale range: 0-24), and self-confidence, comprising items 1, 7, and 9 (subscale range: 0-12).

SECONDARY OUTCOMES:
Patient Dignity Inventory | at baseline assessment before the start of the program and at 3 months immediately after the completion of the study
  The Patient Dignity Inventory (PDI) is a 25-item survey designed to assess dignity-related distress in individuals, particularly those in palliative care. Each item is scored on a 5-point Likert scale, with responses ranging from 1 ("not a problem") to 5 ("an overwhelming problem"). The PDI encompasses five domains of distress: symptom distress, existential distress, dependency, peace of mind, and social support.
Social Frailty Index (SFI) | at baseline assessment before the start of the program and at 3 months immediately after the completion of the study
  The Social Frailty Index (SFI) was developed by Shah et al., 2023, is a multidimensional tool used to evaluate the social aspects of frailty, particularly among older adults. It focuses on identifying individuals at risk of social vulnerabilities that can impact their overall health and well-being. The Social Frailty Index includes age, gender, and eight social characteristics and accurately risk-stratifies older adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Almogama and Dar Alsada assisted living facilities, Damanhur, Damanhur, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after completion of study, the results will be published at data repository platform.